CLINICAL TRIAL: NCT07302425
Title: The Effect of the High-intensity Resistance Training in COPD Patients Recovering From Hospital Exacerbation: a Pilot Study
Brief Title: High-intensity Resistance Training in Post-exacerbation COPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Collaborators: University of Verona, Italy (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICS Maugeri CET6L 0034063/25
Record Dates: First submitted 2025-11-21; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-11

CONDITIONS: COPD Exacerbation
Keywords: COPD; Exacerbation; Early Rehabilitation; High-intensity exercise
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-Intensity Resistance Training (HIRT) (Experimental): This is the group performing high-intensity strength training on the leg press, combined with low-intensity cycling; it is the intervention study group.
  Interventions: Other: HIRT
- High-Intensity Endurance Training (HIET) (Active Comparator): This is the group performing high-intensity endurance training on the cycle ergometer, combined with low-intensity leg press; it is the active comparator study group (Active Comparator).
  Interventions: Other: HIET

INTERVENTIONS:
Other: HIRT — The HIRT group will perform high-intensity strength training on a horizontal leg press, consisting of 4 sets of 5 repetitions at 90-95% of their maximum strength (1RM). Two-minute rests are given between sets, and the weight is increased by 2.5 kg whenever a patient can do more than 5 repetitions. Training focuses on quadriceps strength, from 90° to full extension. Sessions are scheduled 2 days on, 1 day off. This method has been shown to be safe, with mild muscle soreness as the most likely side effect. In addition, participants will perform low-intensity cycling at 20% of their maximum workload, which remains constant throughout the study, to maintain light endurance activity.
  Arms: High-Intensity Resistance Training (HIRT)
Other: HIET — The HIET group will perform high-intensity endurance training on a cycle ergometer for 25 minutes at 70% of their maximum workload, with intensity progression of 10 watts if breathlessness is rated below 5 on the Borg scale. Each session includes a 3-minute warm-up and cool-down, with monitoring of heart rate, blood pressure, oxygen saturation, and symptoms. Participants train 5 days per week. Additionally, they perform low-intensity strength training on the horizontal leg press, 4 sets of 5 repetitions at 20% 1RM, 6-7 days per week, without progression. This combined program maintains both aerobic fitness and light muscle strength during conventional rehabilitation.
  Arms: High-Intensity Endurance Training (HIET)

SUMMARY:
After a COPD exacerbation, many individuals experience severe weakness in the leg muscles, especially the quadriceps. This weakness can make daily activities difficult and slow down recovery. Traditional respiratory rehabilitation usually focuses on endurance training, which is effective but often hard to tolerate soon after an exacerbation due to persistent symptoms and limited functional capacity.

This study aims to compare two early rehabilitation approaches during recovery from a COPD exacerbation: a maximal strength training (MST) programme using high loads and few repetitions, and a traditional endurance-based training programme.

The investigators aim to determine whether MST is easier to tolerate, especially in terms of breathlessness, and whether MST can improve muscle strength, efficiency, and overall exercise tolerance as well as or better than endurance training.

The results will help identify the most suitable rehabilitation strategy for individuals recovering from a COPD exacerbation, particularly for those who struggle with high-intensity endurance exercise.

DETAILED DESCRIPTION:
Background

Exacerbations of chronic obstructive pulmonary disease (COPD) represent critical events in the disease trajectory, significantly increasing mortality, hospital readmissions, and reducing quality of life. Following an exacerbation, affected individuals frequently experience higher symptoms and functional decline, which may be either reversible or not.

Individuals recovering from COPD exacerbations often face profound peripheral muscle weakness, particularly in the quadriceps. This is attributed to systemic inflammation, corticosteroid use, chronic inactivity, and nutritional deficits during acute phases.

Current international guidelines advocate for pulmonary rehabilitation (PR) during the post-acute recovery phase of COPD. These programmes integrate exercise training, self-management education, psychological support, and pharmacological optimization. PR programmes must be tailored to each participant's clinical conditions, comorbidities, and needs.

The ideal timing of PR initiation after an acute exacerbation of COPD remains debated. Some evidence shows that early rehabilitation involving endurance training during hospitalization did not reduce readmission rates nor improve long-term physical capacity, and was associated with increased mortality at 12 months, compared to delayed PR. Consequently, guidelines recommend starting PR within three weeks after discharge from acute hospital care to mitigate any risk associated with early initiation during the acute phase.

Regarding modality, the core component of PR programmes is moderate to high-intensity endurance training, recommended as the gold standard to improve exercise tolerance, functional capacity, and health-related quality of life in stable COPD. However, high-intensity endurance sessions may be hard to tolerate for individuals recovering from an exacerbation, who still experience severe symptoms and marked limitations in daily activities.

Alternative types of training that allow the muscles to be trained without triggering marked dyspnoea and fatigue have been investigated. Previous evidence describes lower cardiorespiratory stress induced by resistance training compared with endurance training in individuals with COPD.

In the context of COPD exacerbations, resistance training initiated early during hospitalization has been shown to effectively prevent muscle deterioration, promote anabolic balance, and counteract catabolic processes without exacerbating systemic inflammation. Individuals undergoing resistance training demonstrated significant improvements in quadriceps strength and six-minute walking distance (6MWD), highlighting its potential as a core component of early PR during COPD exacerbation.

Additional evidence indicates that adding resistance training to endurance training during the post-exacerbation phase produces significant increases in muscle strength while yielding comparable benefits in dyspnoea, exercise capacity, and quality of life.

Therefore, resistance training appears feasible and safe both in the acute and post-acute phases of a COPD exacerbation, but whether strength programmes may allow training for individuals unable to tolerate high-intensity endurance sessions remains unknown.

Among resistance training programmes, maximal strength training (MST) has the potential to most effectively improve lower limb function. MST consists of exercising at high loads and few repetitions, requiring participants to develop maximal rate of force mobilization during the concentric phase. Evidence in stable COPD indicates that MST is safe, feasible, and significantly improves quadriceps rate of force development, mechanical efficiency, and effort tolerance.

Currently, no clear guideline exists for the protocol to be used for participants in the initial rehabilitation phase after exacerbation. In clinical practice, during the early phase of the rehabilitation pathway, a high percentage of individuals (estimated between 40% and 50%) are unable to perform endurance training according to the gold standard for stable COPD (intensity at 70% of maximum watt at incremental test).

For this reason, MST could represent a valid alternative for individuals who are not able or not yet able to tolerate high-intensity endurance training after an exacerbation. Due to the lower respiratory involvement associated with this type of training, the investigators hypothesize higher tolerance, greater improvements in dyspnoea and lower limb muscular efficiency, and similar changes in effort tolerance.

Primary aim

The primary objective of this study is to compare the effects of an early MST programme versus a conventional high-intensity endurance training programme on dyspnoea reduction when initiated shortly after hospital discharge for a COPD exacerbation.

Secondary aims

The secondary aims are to compare MST with high-intensity endurance training in terms of:

1. Functional capacity measured by 6MWD, and exercise tolerance
2. Fatigue reduction over time measured by the Fatigue Severity Scale
3. Muscle strength measured as maximum voluntary contraction of the quadriceps and 1-Repetition Maximum (1RM) on the leg press
4. Impact of the disease and quality of life

   Only for non-dropout participants:
5. Peripheral muscle fatigue assessed through neuromuscular testing
6. Walking efficiency assessed by a dedicated treadmill test

   Only after the last training session:
7. Satisfaction and acceptability of the training programmes

   Material and Methods
   1. Study protocol At enrolment, after providing informed consent, participants will be randomized per block of four by an external operator into two groups (1:1): one group will perform high-intensity resistance training (HIRT, experimental group) and the other conventional endurance training (HIET, control group). Both training programmes will include sessions 5 times/week, of exercises commonly used in respiratory rehabilitation, not involving additional risks compared to normal clinical practice. A senior physiotherapist will supervise all training sessions.
   2. Intervention

      The rehabilitation programme will consist, for the first 15 sessions, of:

   <!-- -->

   1. High-Intensity Resistance Training (HIRT) - Experimental Group Participants will perform high-intensity strength training with progressive workload increases and low-intensity endurance training without progression.

      Strength training will be performed on a horizontal leg press:

      • Four sets of five repetitions at 90-95% of 1RM

      • Focus on concentric quadriceps contraction from 90° to full extension
      * Two-minute rest between sets
      * Load increased by 2.5 kg when participants exceed five repetitions Endurance training will consist of low-intensity cycling at 20% of maximum workload estimated from 6MWD. Intensity will remain unchanged throughout the study.

      Possible side effects include delayed onset muscle soreness (DOMS), typically resolving within a short period.

      HIRT will be performed in cycles of 2 days on and 1 day off.
   2. High-Intensity Endurance Training (HIET) - Control Group

   Participants will perform:

   • Cycling at 70% of maximum workload estimated by 6MWD for 25 minutes

   • Load increased by 10 watts when dyspnoea and fatigue are rated below 5 on the Borg scale
   * Three-minute warm-up and three-minute warm-down
   * Monitoring of heart rate, blood pressure, oxygen saturation, and symptoms at session end
   * Five sessions/week In addition, participants will perform low-intensity resistance training (20% 1RM), four sets of five repetitions on the same leg press, 6-7 days/week, with no progression.

   After the 15-session programme, all participants will undergo T1 evaluation and continue with a combined programme (HIRT + HIET or HIET + HIRT) until discharge.

   3. Dropouts Withdrawal will be defined if participants cannot complete the first training session without adverse events or side effects.

   Criteria:

   - HIRT group: at least 18/20 repetitions completed

   - HIET group: at least 20 minutes of cycling with ≤1-minute interruption Participants unable to complete the first session will be classified as dropouts and continue training at low intensity.

   4. Measures 4.1 Assessments at enrolment

<!-- -->

1. Anthropometric measurements (age, sex, BMI)
2. Comorbidities (CIRS scale)
3. Pulmonary function (spirometry)
4. Arterial blood gases in ambient air

4.2 Outcome measures Collected at T0 (within 3 days of rehabilitation admission), T1 (after 15 sessions), and T2 (discharge).

Primary outcome

• Dyspnoea during daily activities using the Barthel Dyspnoea Index

Secondary outcomes

1. Functional Capacity

   • Six-Minute Walk Test (6MWT): distance, speed, heart rate, oxygen saturation, and Borg dyspnoea/fatigue scores.
2. Fatigue reduction

   * Fatigue Severity Scale (FSS)
3. Muscle Strength and Structure

   • MVC of quadriceps

   • 1RM on horizontal leg press

   • Ultrasound assessment of quadriceps structure

   • Ultrasound assessment of diaphragm structure
4. Disease impact • COPD Assessment Test (CAT) • Maugeri Respiratory Failure 26 (MRF-26) questionnaire

Neuromuscular fatigue (per-protocol only) Assessed using the interpolated twitch technique, including MVC, M waves, electrically stimulated resting force (Qtpot), and maximum voluntary activation (MVA).

Walking efficiency Determined through treadmill test at 3.0 km/h with metabolic analysis.

Acceptability and satisfaction Evaluated after last training session using a Likert scale (0-4).

Sample Size Sample size was calculated based on previous clinical data and expert review, estimating a need for 64 participants (32 per group) to detect meaningful differences in dyspnoea improvement.

Statistical Analysis Data will be analysed using descriptive statistics. Both intention-to-treat and per-protocol analyses will be applied. A two-way repeated-measures ANOVA will assess interaction effects between time (pre/post intervention) and group (resistance vs endurance). Statistical significance is set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* COPD diagnosis according to the GOLD guidelines [11] with FEV1/FVC <70%
* Stable clinical condition (pH>7.30) [11]
* Hospital discharge within 3 weeks from an event of hospitalization due to an acute exacerbation of COPD.
* Absence of significant motor disability, described by the possibility of performing the 6MWT.

Exclusion Criteria:

* Presence of lung diseases other than COPD
* Orthopedic and neurological conditions that prevent the execution of functional tests
* Severe neurological and cardiologic comorbidities or other severe diseases compromise exercise tolerance.
* Cognitive impairment evaluated by Mini-Mental State Examination (MMSE) score as < 25.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-10-30 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Dyspnea during daily activities measured by the Barthel Dyspnea Index (BDI) | From the date of randomization to the End of the program (up to 3 weeks)
  Dyspnea (breathlessness) during routine daily activities will be measured using the Barthel Dyspnea Index (0-100; higher scores indicate greater dyspnea), a questionnaire that evaluates the severity of shortness of breath during common tasks such as walking, dressing, climbing stairs, and bathing. Each activity is scored, and higher scores indicate greater difficulty or breathlessness. The assessment is performed through patient self-report with guidance from a trained clinician. This measure provides a practical evaluation of how dyspnea affects functional independence in everyday life.

SECONDARY OUTCOMES:
Distance walked on the Six-Minute Walk Test (6MWT) | From the date of randomization to the End of the program (up to 3 weeks)
  Distance walked (meters) in the Six-Minute Walk Test (6MWT), measured to assess effort tolerance. The 6MWT evaluates submaximal functional exercise capacity by recording the total distance a patient can walk in six minutes along a flat corridor. It reflects global functional status and endurance.
Fatigue Severity Scale (FSS) total score | From the date of randomization to the End of the program (up to 3 weeks)
  Fatigue severity measured using the Fatigue Severity Scale (FSS; 9 items scored 1-7; higher scores indicate greater fatigue; score range 9 - 63). The FSS assesses the impact of fatigue on daily life and functional performance. Patients rate statements related to fatigue intensity and its effect on physical and social activities.
Maximal Voluntary Contraction (MVC) of isometric quadriceps voluntary strength. | From the date of randomization to the End of the program (up to 3 weeks)
  To evaluate whether HIRT, compared to HIET, increases quadriceps strength, measured as maximal voluntary contraction (MVC) in an isometric leg press position.
Lower Limb Strength Assessment with the 1-Repetition Maximum (1-RM) Test. | From the date of randomization to the End of the program (up to 3 weeks)
  To evaluate whether HIRT, compared to HIET, improves lower-limb strength assessed with the 1-Repetition Maximum (1-RM) test on the horizontal leg press, recording the highest load lifted with rest intervals between trials.
Quadriceps muscle thickness (vastus lateralis) via ultrasound scanning | From the date of randomization to the End of the program (up to 3 weeks)
  Quadriceps (vastus lateralis) muscle thickness, measured in millimeters (mm), assessed via ultrasound imaging. Measurements are taken at standardized anatomical landmarks with participants at rest to evaluate morphological adaptations following the training interventions.
Quadriceps pennation angle (vastus lateralis) via ultrasound scanning | From randomization to the End of the program (up to 3 weeks)
  Quadriceps (vastus lateralis) pennation angle, measured in degrees (°), assessed through ultrasound scanning. Changes in muscle architecture provide insights into structural adaptations associated with training-induced hypertrophy and force-production capacity.
Diaphragmatic thickness via ultrasound scanning | From the date of randomization to the End of the program (up to 3 weeks)
  Diaphragm thickness measured in millimeters (mm) via ultrasound at end-expiration and end-inspiration. This assessment provides insights into structural changes of the diaphragm following the intervention.
Diaphragmatic excursion via ultrasound scanning | From the date of randomization to the End of the program (up to 3 weeks)
  Diaphragmatic excursion, measured in millimeters (mm), assessed via ultrasound during quiet and deep breathing. Excursion reflects diaphragmatic mobility and functional performance.
Impact of the disease (COPD Assessment Test - CAT) | From the date of randomization to the End of the program (up to 3 weeks)
  Disease impact assessed by the COPD Assessment Test (CAT; score 0-40; higher scores indicate worse disease impact). The CAT evaluates symptoms, activity limitations, and overall disease burden from the patient's perspective.
Health-related Quality of Life (MRF-26 questionnaire) | From the date of randomization to the End of the program (up to 3 weeks)
  Health-related quality of life evaluated using the Maugeri Respiratory Failure 26 questionnaire (MRF-26; score 0-78; higher scores indicate worse quality of life). The questionnaire focuses on physical function, disability, and respiratory-related limitations..
Maximal Voluntary Contraction (MVC) | From the date of randomization to the End of the program (up to 3 weeks)
  Maximal Voluntary Contraction (MVC), measured Newtons (N), before and after the standardized fatigue task using dynamometry to quantify voluntary quadriceps force production.
Electrically stimulated resting force (Qtpot) | From the date of randomization to the End of the program (up to 3 weeks)
  Electrically stimulated potentiated twitch force (Qtpot), measured in Newtons (N), used to assess peripheral muscle fatigue and contractile function.
Maximal Voluntary Activation (MVA) | From the date of randomization to the End of the program (up to 3 weeks)
  Maximal voluntary activation (%) assessed via the interpolated twitch technique, quantifying central drive and central fatigue.
M-wave amplitude | From the date of randomization to the End of the program (up to 3 weeks)
  M-wave amplitude recorded through surface electromyography (EMG) and measured in millivolts (mV), to evaluate neuromuscular transmission and peripheral excitability before and after the fatigue task.
Walking efficiency (Walking Energy cost). | From the date of randomization to the End of the program (up to 3 weeks)
  To evaluate whether HIRT, compared to HIET, improves walking efficiency, measured as the energy cost of walking on a treadmill for six minutes at 3 km/h, using oxygen consumption data collected via a portable metabolic analyzer.
Acceptability and satisfaction with the training. | From the date of randomization to the End of the program (up to 3 weeks)
  To evaluate the acceptability and satisfaction of participants with the training programs, assessed using a Likert scale from 0 (completely unsatisfied) to 4 (very high satisfaction) after the last training session.

CONTACTS AND LOCATIONS:
Overall Officials: Mara Paneroni, PhD, MSc, Study Director — ICS Maugeri IRCCS, respiratory rehabilitation of the Institute of Lumezzane
Locations (1):
- ICS Maugeri IRCCS, Respiratory rehabilitation of the Institute of Lumezzane, Lumezzane, Brescia, Italy

REFERENCES:
- [Background] Vitacca M, Malovini A, Paneroni M, Spanevello A, Ceriana P, Capelli A, Murgia R, Ambrosino N. Predicting Response to In-Hospital Pulmonary Rehabilitation in Individuals Recovering From Exacerbations of Chronic Obstructive Pulmonary Disease. Arch Bronconeumol. 2024 Mar;60(3):153-160. doi: 10.1016/j.arbres.2024.01.001. Epub 2024 Jan 17. English, Spanish. PMID 38296674
- [Background] Norman G. Likert scales, levels of measurement and the "laws" of statistics. Adv Health Sci Educ Theory Pract. 2010 Dec;15(5):625-32. doi: 10.1007/s10459-010-9222-y. Epub 2010 Feb 10. PMID 20146096
- [Background] Gaesser GA, Brooks GA. Muscular efficiency during steady-rate exercise: effects of speed and work rate. J Appl Physiol. 1975 Jun;38(6):1132-9. doi: 10.1152/jappl.1975.38.6.1132. PMID 1141128
- [Background] Amann M, Romer LM, Subudhi AW, Pegelow DF, Dempsey JA. Severity of arterial hypoxaemia affects the relative contributions of peripheral muscle fatigue to exercise performance in healthy humans. J Physiol. 2007 May 15;581(Pt 1):389-403. doi: 10.1113/jphysiol.2007.129700. Epub 2007 Feb 22. PMID 17317739
- [Background] Vidotto G, Carone M, Jones PW, Salini S, Bertolotti G; Quess Group. Maugeri Respiratory Failure questionnaire reduced form: a method for improving the questionnaire using the Rasch model. Disabil Rehabil. 2007 Jul 15;29(13):991-8. doi: 10.1080/09638280600926678. PMID 17612984
- [Background] Dal Negro RW, Bonadiman L, Turco P. Sensitivity of the COPD assessment test (CAT questionnaire) investigated in a population of 681 consecutive patients referring to a lung clinic: the first Italian specific study. Multidiscip Respir Med. 2014 Mar 15;9(1):15. doi: 10.1186/2049-6958-9-15. PMID 24629022
- [Background] Jia Y, Zhang Q. Research Progress on Diaphragm Ultrasound in Chronic Obstructive Pulmonary Disease: A Narrative Review. Ultrasound Med Biol. 2022 Apr;48(4):587-597. doi: 10.1016/j.ultrasmedbio.2021.10.019. Epub 2022 Jan 19. PMID 35065813
- [Background] Ottonello M, Pellicciari L, Giordano A, Foti C. Rasch analysis of the Fatigue Severity Scale in Italian subjects with multiple sclerosis. J Rehabil Med. 2016 Jul 18;48(7):597-603. doi: 10.2340/16501977-2116. PMID 27344968
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Vitacca M, Malovini A, Balbi B, Aliani M, Cirio S, Spanevello A, Fracchia C, Maniscalco M, Corica G, Ambrosino N, Paneroni M. Minimal Clinically Important Difference in Barthel Index Dyspnea in Patients with COPD. Int J Chron Obstruct Pulmon Dis. 2020 Oct 21;15:2591-2599. doi: 10.2147/COPD.S266243. eCollection 2020. PMID 33116476
- [Background] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Background] Salvi F, Miller MD, Grilli A, Giorgi R, Towers AL, Morichi V, Spazzafumo L, Mancinelli L, Espinosa E, Rappelli A, Dessi-Fulgheri P. A manual of guidelines to score the modified cumulative illness rating scale and its validation in acute hospitalized elderly patients. J Am Geriatr Soc. 2008 Oct;56(10):1926-31. doi: 10.1111/j.1532-5415.2008.01935.x. Epub 2008 Sep 22. PMID 18811613
- [Background] Luxton N, Alison JA, Wu J, Mackey MG. Relationship between field walking tests and incremental cycle ergometry in COPD. Respirology. 2008 Nov;13(6):856-62. doi: 10.1111/j.1440-1843.2008.01355.x. PMID 18811884
- [Background] Cheung K, Hume P, Maxwell L. Delayed onset muscle soreness : treatment strategies and performance factors. Sports Med. 2003;33(2):145-64. doi: 10.2165/00007256-200333020-00005. PMID 12617692
- [Background] Global Initiative for Chronic Obstructive Lung Disease (GOLD) Global Strategy for Prevention, Diagnosis and Management of COPD: 2024 Report. Bethesda: GOLD; https://goldcopd.org/2024-gold-report
- [Background] Hoff J, Tjonna AE, Steinshamn S, Hoydal M, Richardson RS, Helgerud J. Maximal strength training of the legs in COPD: a therapy for mechanical inefficiency. Med Sci Sports Exerc. 2007 Feb;39(2):220-6. doi: 10.1249/01.mss.0000246989.48729.39. PMID 17277584
- [Background] Daabis R, Hassan M, Zidan M. Endurance and strength training in pulmonary rehabilitation for COPD patients. Egypt J Chest Dis Tuberc. 2017;66(2):231-236. doi:10.1016/j.ejcdt.2016.07.003
- [Background] Troosters T, Probst VS, Crul T, Pitta F, Gayan-Ramirez G, Decramer M, Gosselink R. Resistance training prevents deterioration in quadriceps muscle function during acute exacerbations of chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2010 May 15;181(10):1072-7. doi: 10.1164/rccm.200908-1203OC. Epub 2010 Feb 4. PMID 20133927
- [Background] Probst VS, Troosters T, Pitta F, Decramer M, Gosselink R. Cardiopulmonary stress during exercise training in patients with COPD. Eur Respir J. 2006 Jun;27(6):1110-8. doi: 10.1183/09031936.06.00110605. Epub 2006 Mar 15. PMID 16540501
- [Background] Greening NJ, Williams JE, Hussain SF, Harvey-Dunstan TC, Bankart MJ, Chaplin EJ, Vincent EE, Chimera R, Morgan MD, Singh SJ, Steiner MC. An early rehabilitation intervention to enhance recovery during hospital admission for an exacerbation of chronic respiratory disease: randomised controlled trial. BMJ. 2014 Jul 8;349:g4315. doi: 10.1136/bmj.g4315. PMID 25004917
- [Background] Spruit MA, Singh SJ, Garvey C, ZuWallack R, Nici L, Rochester C, Hill K, Holland AE, Lareau SC, Man WD, Pitta F, Sewell L, Raskin J, Bourbeau J, Crouch R, Franssen FM, Casaburi R, Vercoulen JH, Vogiatzis I, Gosselink R, Clini EM, Effing TW, Maltais F, van der Palen J, Troosters T, Janssen DJ, Collins E, Garcia-Aymerich J, Brooks D, Fahy BF, Puhan MA, Hoogendoorn M, Garrod R, Schols AM, Carlin B, Benzo R, Meek P, Morgan M, Rutten-van Molken MP, Ries AL, Make B, Goldstein RS, Dowson CA, Brozek JL, Donner CF, Wouters EF; ATS/ERS Task Force on Pulmonary Rehabilitation. An official American Thoracic Society/European Respiratory Society statement: key concepts and advances in pulmonary rehabilitation. Am J Respir Crit Care Med. 2013 Oct 15;188(8):e13-64. doi: 10.1164/rccm.201309-1634ST. PMID 24127811
- [Background] Polkey MI. Peripheral muscle weakness in COPD: where does it come from? Thorax. 2003 Sep;58(9):741-2. doi: 10.1136/thorax.58.9.741. No abstract available. PMID 12947126
- [Background] Abdulai RM, Jensen TJ, Patel NR, Polkey MI, Jansson P, Celli BR, Rennard SI. Deterioration of Limb Muscle Function during Acute Exacerbation of Chronic Obstructive Pulmonary Disease. Am J Respir Crit Care Med. 2018 Feb 15;197(4):433-449. doi: 10.1164/rccm.201703-0615CI. PMID 29064260
- [Background] Pitta F, Troosters T, Probst VS, Spruit MA, Decramer M, Gosselink R. Physical activity and hospitalization for exacerbation of COPD. Chest. 2006 Mar;129(3):536-44. doi: 10.1378/chest.129.3.536. PMID 16537849
- [Background] Wedzicha JA Ers Co-Chair, Miravitlles M, Hurst JR, Calverley PM, Albert RK, Anzueto A, Criner GJ, Papi A, Rabe KF, Rigau D, Sliwinski P, Tonia T, Vestbo J, Wilson KC, Krishnan JA Ats Co-Chair. Management of COPD exacerbations: a European Respiratory Society/American Thoracic Society guideline. Eur Respir J. 2017 Mar 15;49(3):1600791. doi: 10.1183/13993003.00791-2016. Print 2017 Mar. PMID 28298398